CLINICAL TRIAL: NCT05267470
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Bemarituzumab Monotherapy and Combination With Other Anti-Cancer Therapy in Subjects With Squamous-Cell Non-Small-Cell Lung Cancer (FORTITUDE-201)
Brief Title: A Study of Bemarituzumab Monotherapy and Combination With Other Anti-cancer Therapy in SqNSCLC With FGFR2b Overexpression (FORTITUDE-201)
Acronym: FORTITUDE-201
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision not due to safety concerns
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20210102; 2021-004058-47 (EudraCT Number); 2023-505456-22 (Other: EU CT Number)
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Squamous-Cell Non-Small-Cell Lung Cancer
Keywords: Squamous-Cell Non-Small-Cell Lung Cancer; FGFR2b-positive Squamous-Cell Non-Small-Cell Lung Cancer; SqNSCLC; Bemarituzumab; Docetaxel
MeSH Terms: interventions — bemarituzumab; Docetaxel; pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Combination Dose Exploration (Experimental): Participants with SqNSCLC will receive escalating doses of bemarituzumab in combination with docetaxel.
  Interventions: Drug: Bemarituzumab; Drug: Docetaxel
- Part 2: Combination Dose Expansion (Experimental): Participants with SqNSCLC and FGFR2b overexpression will receive the dose of bemarituzumab in combination with docetaxel identified as safe during Part 1.
  Interventions: Drug: Bemarituzumab; Drug: Docetaxel
- Part 3: Bemarituzumab Monotherapy (Experimental): Participants with SqNSCLC and FGFR2b overexpression will receive bemarituzumab monotherapy.
  Interventions: Drug: Bemarituzumab
- Part 4: Combination Immuno-chemotherapy (Experimental): Participants with FGFR2b overexpression will receive the dose of bemarituzumab identified as safe during Part 1 in combination with pembrolizumab, carboplatin and either paclitaxel or nab-paclitaxel.
  Interventions: Drug: Bemarituzumab; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Bemarituzumab — Intravenous (IV) infusion
  Other Names: AMG 552
Drug: Docetaxel — IV infusion
  Arms: Part 1: Combination Dose Exploration; Part 2: Combination Dose Expansion
Drug: Pembrolizumab — IV infusion
  Arms: Part 4: Combination Immuno-chemotherapy
Drug: Carboplatin — IV infusion
  Arms: Part 4: Combination Immuno-chemotherapy
Drug: Paclitaxel — IV infusion
  Arms: Part 4: Combination Immuno-chemotherapy
Drug: Nab-paclitaxel — IV infusion
  Arms: Part 4: Combination Immuno-chemotherapy

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of bemarituzumab monotherapy and combination with other anti-cancer therapies, and to determine the recommended phase 3 dose of bemarituzumab in combination with other anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures
* Age ≥ 18 years old (or legal adult within country, whichever is older) at the time that the Informed Consent Form (ICF) is signed
* Pathologically confirmed squamous cell lung carcinoma
* Disease that is unresectable, locally advanced or metastatic (not amenable to curative therapy)
* Participants must have archived tumor tissue sample (formalin fixed, paraffin embedded [FFPE] sample [FFPE of excisional, or core needle]) taken within last 5 years or be willing to undergo pre-treatment tumor biopsy (excisional, or core needle) for tissue prior to enrollment
* Participant must have progressed on, or recurred after at least 1 prior systemic therapy (Part 1 and 2 only) or at least 2 prior systemic therapies (Part 3 only) for locally advanced and unresectable or metastatic disease. Prior treatment must include a platinum-based doublet chemotherapy and checkpoint inhibitor for advanced or metastatic disease, either given as one line of therapy or as individual lines of therapy, unless the participant has a medical contraindication to one of the required therapies (which must be documented in the electronic case report form [eCRF]). Additionally, if the participant's tumor was previously identified as having a driver mutation (according to local standard of care or guidelines, e.g., Kirsten rat sarcoma [KRAS] G12C, neurotrophic tyrosine receptor kinase [NTRK]), which has an approved therapy for which the participant is eligible and available, the participant must have received the approved therapy in a prior line of treatment.
* For Part 4, participants may not have received prior systemic therapy for their locally advanced and unresectable or metastatic disease. For Part 4, participants who received peri-operative systemic therapy are eligible if that adjuvant/neoadjuvant therapy was completed at least 12 months prior to diagnosis of locally advanced and unresectable or metastatic disease.
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function as determined per protocol
* Part 2, 3 and 4 only: FGFR2b overexpression as determined by centrally performed immunohistochemistry (IHC) testing

Exclusion Criteria:

* Mixed small-cell lung cancer or mixed non-small cell lung cancer (NSCLC) histology
* Untreated or symptomatic central nervous system (CNS) metastases or leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures at a frequency greater than monthly
* Impaired cardiac function or clinically significant cardiac disease including: unstable angina within 6 months prior to first dose of study treatment, acute myocardial infarction < 6 months prior to first dose of study treatment, New York Heart Association (NYHA) class II-IV congestive heart failure, uncontrolled hypertension (defined as an average systolic blood pressure >160 mmHg or diastolic >100 mm Hg despite optimal treatment (measured following European Society for Hypertension/European Society of Cardiology [ESH/ESC] 2013 guidelines; Section 11.11), uncontrolled cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, active coronary artery disease, Fridericia's correction formula (QTc) ≥ 470
* Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks) or actively progressing
* Recent (within 6 months) corneal surgery or ophthalmic laser treatment or recent (within 6 months) history of, or evidence of, corneal defects, corneal ulcerations, keratitis, or keratoconus, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer
* Part 1 and Part 2: participants that experienced toxicity or hypersensitivity requiring discontinuation of prior docetaxel treatment
* Part 1 only: participants that had disease progression on prior therapy with docetaxel
* Part 2 only: participants have received prior docetaxel in unresectable or metastatic setting (including participants who received prior docetaxel in first line for metastatic disease, but not including participants who received prior docetaxel neoadjuvantly or adjuvantly and did not progress within 6 months of end of therapy)
* Prior treatment with any selective inhibitor of the fibroblast growth factor-fibroblast growth factor receptor (FGF-FGFR) pathway

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (39):
- United States (4):
  - University of California Irvine, Orange, California
  - Morristown Medical Center, Morristown, New Jersey
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University of Pittsburgh, Cancer Institute, Pittsburgh, Pennsylvania
- Belgium (4):
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
- France (6):
  - Institut Bergonie, Bordeaux
  - CHU de Lyon - Hopital Louis Pradel, Bron
  - Hôpital Tenon, Paris
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Institut Gustave Roussy, Villejuif
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Poland (7):
  - Przychodnia Lekarska Komed Roman Karaszewski, Konin
  - Pratia Mcm Krakow, Krakow
  - Krakowskie Centrum Medyczne Sp zoo, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Instytut Genetyki i Immunologii GENIM Spzoo, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Mazowieckie centrum leczenia, Otwock
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (9):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet. Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Complexo Hospitalario Universitario A Coruña Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 participants were enrolled across 8 countries from March 2022 and the last participant last visit was in May 2024.
Pre-assignment Details: The study consisted of 4 Parts:
  * Part 1: Combination dose exploration with docetaxel
  * Part 2: Combination dose expansion with docetaxel
  * Part 3: Monotherapy
  * Part 4: Combination with carboplatin, paclitaxel or nab-paclitaxel, and pembrolizumab.
  The planned dose levels were dose level 1 (lower) and dose level 2 (higher).
Groups:
- Part 1: Bemarituzumab Dose 1 With Docetaxel: Participants received multiple intravenous (IV) doses of bemarituzumab dose level 1 and IV docetaxel (cycle length = 21 days).
- Part 1: Bemarituzumab Dose 2 With Docetaxel: Participants received multiple IV doses of bemarituzumab dose level 2 and IV docetaxel (cycle length = 21 days).
- Part 2: Bemarituzumab Dose 2 With Docetaxel: Participants who had an overexpression of FGFR2b received multiple IV doses of bemarituzumab dose level 2 and IV docetaxel (cycle length = 21 days).
- Part 3: Bemarituzumab Dose 1: Participants who had an overexpression of FGFR2b received multiple IV doses of bemarituzumab dose level 1 (cycle length = 14 days).
- Part 4: Bemarituzumab Dose 2 First-line Combination Therapy: Participants who had an overexpression of FGFR2b received multiple IV doses of bemarituzumab dose level 2 in combination with pembrolizumab, carboplatin and either paclitaxel or nab-paclitaxel (cycle length = 21 days).
Period: Overall Study
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Started | 4 | 9 | 29 | 28 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 29 | 28 | 4
Not completed — Decision by sponsor | 0 | 3 | 19 | 7 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2 | 0
Not completed — Death | 3 | 5 | 8 | 18 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Bemarituzumab Dose 1 With Docetaxel: Participants received multiple IV doses of bemarituzumab dose level 1 and IV docetaxel (cycle length = 21 days).
- Total: Total of all reporting groups
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy | Total
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (4.5) | 65.9 (8.5) | 65.3 (6.2) | 63.0 (8.2) | 63.0 (7.9) | 64.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 8 | 0 | 12
  Male | 4 | 7 | 27 | 20 | 4 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 9 | 27 | 27 | 4 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 4 | 12 | 12 | 3 | 33
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 2 | 4 | 14 | 11 | 1 | 32
  Other | 0 | 0 | 1 | 0 | 0 | 1
  Missing | 0 | 1 | 1 | 5 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT): Parts 1 and 4
Description: DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and included the below if considered by the investigator to be related to study drug, excluding toxicities related to disease progression or intercurrent illness: Grade 3 thrombocytopenia for > 7 days or with Grade > 2 bleeding, vomiting/diarrhea for > 3 days, fatigue; Grade ≥ 3 febrile neutropenia, nausea for > 3 days; Grade 4 neutropenia, thrombocytopenia, anemia, ophthalmologic AE, laboratory value, vomiting/diarrhea; Grade 5 toxicity (death not due to disease progression). CTCAE Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, and Grade 5 results in death.
Time Frame: Day 1 to Day 21 of Cycle 1 (each cycle was 21 days)
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 4
Participants | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participants. TEAEs were any AE that started on or after receiving the first dose of investigational product and up to 28 days after the last dose of investigational product or the end of study date, whichever is earlier. Treatment-related TEAEs were those considered possibly related to study treatment by the investigator. Any clinically significant changes in electrocardiograms, vital signs, physical examination with a neurological assessment, clinical laboratory tests, and visual acuity were recorded as TEAEs. A serious TEAE resulted in death, was immediately life threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event. AEs of special interest (AESIs) were ocular events of any CTCAE grade or seriousness occurring up to 100 days after the last dose of bemarituzumab.
Time Frame: Day 1 of cycle 1 to 100 days after the last dose of study treatment or end of study date, whichever occurred earlier (Parts 1, 2, and 4 cycle length = 21 days; Part 3 cycle length = 14 days). Median treatment duration was 6.2 weeks.
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4
Participants
  Any TEAE | 4 | 9 | 29 | 25 | 4
  Any SAE | 4 | 5 | 16 | 8 | 4
  Any treatment-related TEAE | 3 | 9 | 21 | 16 | 2
  Any treatment-related SAE | 0 | 0 | 2 | 0 | 2
  Any AESI | 2 | 6 | 17 | 9 | 2

3. Secondary Outcome: Area Under the Serum Drug Concentration-time Curve From Time 0 to End of Dosing Interval (AUCtau) of Bemarituzumab
Description: Bemarituzumab serum concentrations with values below the limit of quantification were set to zero for analysis. Pharmacokinetic (PK) parameters were determined from the time concentration profile using noncompartmental analysis.
Time Frame: Parts 1, 2, 3, and 4: Cycles 1 and 2 pre-dose, 0.25, 3, 6, 24, 72, 168, 336, 504 (except Part 3) hours post-dose
Population: The PK analysis set included all participants who received at least one dose of bemarituzumab and had at least one PK sample collected. Participants with data available at each timepoint are presented.
Measure: Median (Full Range); unit: day*mcg/mL
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 25 | 3
day*mcg/mL
  Cycle 1: number analyzed (Participants) | 4 | 8 | 29 | 24 | 3
  Cycle 1 | 3370 [2400 to 4880] | 5300 [3830 to 6870] | 3920 [2290 to 6470] | 2800 [1360 to 4820] | 3020 [2000 to 3270]
  Cycle 2: number analyzed (Participants) | 3 | 9 | 21 | 25 | 2
  Cycle 2 | 2610 [2160 to 4810] | 4850 [1190 to 7290] | 4000 [1200 to 10300] | 3580 [1880 to 5970] | 2340 [1470 to 3200]

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Bemarituzumab
Description: Bemarituzumab serum concentrations with values below the limit of quantification were set to zero for analysis. PK parameters were determined from the time concentration profile using noncompartmental analysis.
Time Frame: Parts 1, 2, 3, and 4: Cycles 1 and 2 pre-dose, 0.25, 3, 6, 24, 72, 168, 336, 504 (except Part 3) hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 25 | 3
mcg/mL
  Cycle 1 | 599 [457 to 751] | 746 [627 to 896] | 646 [338 to 956] | 398 [238 to 1430] | 561 [463 to 564]
  Cycle 2: number analyzed (Participants) | 3 | 9 | 21 | 25 | 2
  Cycle 2 | 379 [358 to 599] | 715 [595 to 910] | 601 [314 to 845] | 532 [314 to 811] | 322 [235 to 409]

5. Secondary Outcome: Observed Concentration at the End of a Dose Interval (Ctrough) of Bemarituzumab
Description: as for outcome 4
Time Frame: Pre-dose Cycle 2 Day 1 and Cycle 3 day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 3 | 9 | 21 | 26 | 3
mcg/mL
  Pre-dose Cycle 2 Day 1 | 51.5 [25.8 to 96.6] | 93.7 [40.2 to 175] | 88.9 [50.5 to 154] | 147 [10.1 to 554] | 29.9 [25.3 to 32.5]
  Pre-dose Cycle 3 Day 1: number analyzed (Participants) | 3 | 6 | 13 | 25 | 1
  Pre-dose Cycle 3 Day 1 | 79.1 [33.9 to 112] | 149 [45.0 to 201] | 111 [30.6 to 169] | 140 [29.3 to 271] | 69.2 [69.2 to 69.2]

6. Secondary Outcome: Percentage of Participants Who Achieved an Objective Response (OR)
Description: OR was defined as the best overall response of confirmed complete response (CR) or confirmed partial response (PR) as defined by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. All lymph nodes must have been non-pathological in size (< 10 mm).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 6 (+/- 1) weeks from the first dose of bemarituzumab (cycle 1 day 1) up to week 54, then every 12 (+/- 2 weeks), up to the end of the long term follow-up (LTFU) period (median time on study was approximately 21 weeks)
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4
percentage of participants | 0.0 [0.0 to 60.2] | 22.2 [2.8 to 60.0] | 10.3 [2.2 to 27.4] | 0.0 [0.0 to 12.3] | 25.0 [0.6 to 80.6]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of OR (determined by the investigator per RECIST v1.1) until first documentation of disease progression or death due to any cause, whichever occurred first.
  DOR was censored at the last evaluable post-baseline tumor assessment prior to subsequent anticancer therapy; otherwise, at date of first documentation of OR (i.e., assigned a one-day interval).
Time Frame: Every 6 (+/- 1) weeks from the first dose of bemarituzumab (cycle 1 day 1) up to week 54, then every 12 (+/- 2 weeks), up to the end of the LTFU period (median time on study was approximately 21 weeks)
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab. Only participants who had achieved OR were evaluated for DOR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 0 | 2 | 3 | 0 | 1
months |  | 5.5 [2.8 to NA] — Upper confidence interval (CI) was not calculable due to insufficient event data occurring above the median. | 2.8 [2.8 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. |  | 4.5 [NA to NA] — CIs were not calculable due to only 1 participant achieving OR.

8. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants documented to have a CR, PR or stable disease (SD) per RECIST v1.1.
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to <10 mm. All lymph nodes must have been non-pathological in size (< 10 mm).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5 mm. Unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 7
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4
percentage of participants | 75.0 [19.4 to 99.4] | 66.7 [29.9 to 92.5] | 65.5 [45.7 to 82.1] | 53.6 [33.9 to 72.5] | 75.0 [19.4 to 99.4]

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from date of first dose of investigational product until the first documentation of radiologic disease progression or death due to any cause, whichever occurred first, in the absence of subsequent anticancer therapy.
  PFS was censored at the last evaluable post-baseline tumor assessment prior to subsequent anticancer therapy; otherwise, at first dose of investigational product. Progression was based on RECIST v1.1 criteria.
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5 mm. Unequivocal progression of existing non-target lesions.
Time Frame: Participants completed the LTFU for survival every 3 months ± 1 month after the safety follow-up visit (at 28 days after the last dose of bemarituzumab), up to the end of the study. Median time on study was approximately 21 weeks
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4
months | 4.2 [1.2 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 4.2 [1.4 to 10.8] | 4.0 [1.4 to 4.4] | 1.8 [1.3 to 2.6] | 5.6 [1.3 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of investigational product until event of death due to any cause through the analysis cutoff date. Participants still alive were censored at the date last known to be alive through the analysis cutoff date.
Time Frame: as for outcome 9
Population: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
Number analyzed (Participants) | 4 | 9 | 29 | 28 | 4
months | 6.0 [5.6 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 12.8 [3.3 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | NA [9.1 to NA] — Median and upper CI were not calculable due to fewer than 50% events. | 5.4 [2.8 to 8.0] | NA [3.5 to NA] — Median and upper CI were not calculable due to fewer than 50% events.

ADVERSE EVENTS:
Time Frame: For all cause mortality, from first dose of bemarituzumab until end of study; median (min, max) time on study was 20.79 [1.9, 83.7] weeks. For serious AEs and other AEs, Day 1 of cycle 1 to 100 days after the last dose of study treatment or end of study date, whichever occurred earlier (Parts 1, 2, and 4 cycle length = 21 days; Part 3 cycle length = 14 days). Median treatment duration was 6.2 weeks.
Description: The safety analysis set included all participants who received at least one dose of bemarituzumab.
Arm/Group | Part 1: Bemarituzumab Dose 1 With Docetaxel | Part 1: Bemarituzumab Dose 2 With Docetaxel | Part 2: Bemarituzumab Dose 2 With Docetaxel | Part 3: Bemarituzumab Dose 1 | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy
All-Cause Mortality (participants affected / at risk) | 3/4 | 5/9 | 8/29 | 18/28 | 1/4
Serious Adverse Events (participants affected / at risk) | 4/4 | 5/9 | 16/29 | 8/28 | 4/4
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 26/29 | 23/28 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Bemarituzumab Dose 1 With Docetaxel (N=4) | Part 1: Bemarituzumab Dose 2 With Docetaxel (N=9) | Part 2: Bemarituzumab Dose 2 With Docetaxel (N=29) | Part 3: Bemarituzumab Dose 1 (N=28) | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericarditis malignant (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Corneal epithelium defect (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Cerebral disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Bemarituzumab Dose 1 With Docetaxel (N=4) | Part 1: Bemarituzumab Dose 2 With Docetaxel (N=9) | Part 2: Bemarituzumab Dose 2 With Docetaxel (N=29) | Part 3: Bemarituzumab Dose 1 (N=28) | Part 4: Bemarituzumab Dose 2 First-line Combination Therapy (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 6 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 5 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Acute macular neuroretinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 5 | 3 | 0
Cataract (Eye disorders) | 1 | 1 | 1 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 2 | 1 | 0
Corneal disorder (Eye disorders) | 1 | 3 | 2 | 2 | 1
Corneal epithelium defect (Eye disorders) | 0 | 1 | 3 | 0 | 1
Corneal opacity (Eye disorders) | 0 | 1 | 0 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 2 | 4 | 0
Keratitis (Eye disorders) | 0 | 0 | 3 | 0 | 0
Keratopathy (Eye disorders) | 1 | 2 | 10 | 4 | 0
Limbal stem cell deficiency (Eye disorders) | 0 | 1 | 4 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 1 | 0 | 1
Retinal drusen (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 1 | 0
Visual acuity reduced (Eye disorders) | 3 | 6 | 15 | 9 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 8 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 4 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 10 | 2 | 1
Fatigue (General disorders) | 0 | 2 | 1 | 3 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 4 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 3 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 8 | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT05267470/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05267470/SAP_001.pdf